CLINICAL TRIAL: NCT03250546
Title: Randomized Prospective Phase II Clinical Trial Using Post-Transplantation Cyclophosphamide for Prevention of GVHD in Haploidentical and HLA-9/10 Mismatched Unrelated Donors Hematopoietic Stem Cell Transplant
Brief Title: Haploidentical and Mismatched Unrelated Donors Hematopoietic Stem Cell Transplant
Acronym: ALTERGREF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P151001
Record Dates: First submitted 2017-07-31; First posted 2017-08-15 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Hematopoietic Stem Cell Transplant

STUDY DESIGN:
Intervention Model Description: Randomized prospective Phase II Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haplo-identical group (Experimental)
  Interventions: Procedure: transplant from a haplo-identical donor
- HLA-9/10 MMUD group (Active Comparator)
  Interventions: Procedure: transplant from a non related donor

INTERVENTIONS:
Procedure: transplant from a haplo-identical donor — The transplant procedures will be similar in the 2 groups beside the origin of cells
  Arms: Haplo-identical group
Procedure: transplant from a non related donor — The transplant procedures will be similar in the 2 groups beside the origin of cells
  Arms: HLA-9/10 MMUD group

SUMMARY:
The primary objective of this study is to compare the 2-year progression free survival without acute graft versus host disease (GvHD) (aGvHD) grade III-IV or without moderate or severe chronic (cGVHD) after transplant from haploidentical hematopoietic stell cell transplant (HSCT) or from an unrelated Human Leukocyte Antigen (HLA)-9/10 mismatched unrelated donor (MMUD).

It will use a Phase II, multicenter, prospective, randomized clinical trial.

By setting a power of 80% and a type I error rate of 5% for a two-sided log-rank test (hypotheses tested: probability of event-free survival at 2 years 50% vs. 30 %), 92 patients need to be recruited in each arm, for a total of 184 patients.

ELIGIBILITY:
Inclusion Criteria:

* With a hematological malignancy requiring a HSCT and at least in partial response ie a) Acute Leukemia in complete remission, b) Myelodysplastic syndromes with less than 20% marrow, c) Myeloproliferative syndromes with less than 20% bone marrow blasts, d) Non Hodgkin Lymphoma (NHL), Hodgkin's disease, chronic lymphocytic leukemia at least in partial response, e) Myeloma at least in partial response.
* Without HLA matched related or unrelated donor
* Identification of a possible HLA-9/10 MMUD and a possible haplo-identical donor.
* Having read and understood the information letter and signed the informed consent
* With health insurance coverage

Exclusion Criteria:

* Organic or psychiatric disease, non related to the hematological malignancy, contraindicating the transplant.
* Performance Scale by the Eastern Cooperative Oncology Group (ECOG)> 2
* Severe uncontrolled infection
* Cardiac contraindication of post-transplant Cy (coronary insufficiency, ejection ventricular fraction <50%)
* Aspartate transaminase (AST) and alanine transaminase (ALT) > 2.5 N, creatinine > 150 mmol/L (except if related to malignancy)
* Previous active cancer in the last two years, except basal cell skin cancer and in situ carcinoma of the cervix
* Childbearing age woman refusing contraception
* Patients who did not accept the follow-up planned by the protocol
* Positive serology for HIV or Human T-Lymphotropic Virus (HTLV)-1, 2, or active viral infection by the Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV)
* Pregnant woman (positive β-HCG) or during lactation
* Adult patient on guardianship, or safeguard justice

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Two-year progression free survival, without acute GVHD grade III-IV and without moderate/severe cGVHD | 2 year

SECONDARY OUTCOMES:
100 day engraftment | day 100

OTHER OUTCOMES:
Overall survival | 2 year
Progression Free survival | 2 year
Cumulative incidence of progression | 2 year
Acute GVHD incidence | day 100
Chronic GVHD incidence | 2 year
Non relapse Mortality (NRM) | year 2
Stages of Chimerism | month 1, 2, 3, 6 and 12
  * Complete chimerism: 100% donor cells detected, suggesting complete hematopoietic replacement
  * Mixed chimerism: Host cells are detected in particular cells like lymphocytes. Five to 90% donor cells
  * Split chimerism: One or more lineages are of host and one or more lineages are of donor, like myeloid cells are 100% host and T-cells are 100% donor.
Severe infections | 2 year
Time interval between diagnosis and transplant | day 100
Adverse events | day 100 and two years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Saint Louis hospital, Paris
  - Service Hématologie Clinique, Paris